CLINICAL TRIAL: NCT01058005
Title: A Multicenter, Randomized, Open-Label, Parallel-Group, Active-Controlled Study to Evaluate the Benefits of Switching Therapy (Glatiramer Acetate or Interferon Beta-1a) to Natalizumab in Subjects With Relapsing Remitting Multiple Sclerosis
Brief Title: Study Evaluating Rebif, Copaxone, and Tysabri for Active Multiple Sclerosis
Acronym: SURPASS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to significantly slower than expected enrollment, the Sponsor decided to terminate the study.
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 101MS325
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab; Interferon beta-1a; Glatiramer Acetate

ARMS (3):
- Natalizumab (Experimental)
  Interventions: Drug: BG00002 (natalizumab)
- Interferon Beta-1a (Active Comparator)
  Interventions: Drug: interferon beta-1a
- Glatiramer Acetate (Active Comparator)
  Interventions: Drug: glatiramer acetate

INTERVENTIONS:
Drug: BG00002 (natalizumab) — 300 mg intravenous injection every 4 weeks
  Other Names: Tysabri
  Arms: Natalizumab
Drug: interferon beta-1a — 44 mcg subcutaneous injection 3 times per week
  Other Names: Rebif
  Arms: Interferon Beta-1a
Drug: glatiramer acetate — 20 mg subcutaneous injection once daily
  Other Names: Copaxone
  Arms: Glatiramer Acetate

SUMMARY:
This was a multicenter, randomized, open-label, parallel-group, active-controlled study. Prior to randomization, participants were to have been treated with glatiramer acetate or interferon β-1a (44 μg). Participants were to be randomized to receive natalizumab, interferon β-1a 44 μg, or glatiramer acetate.

DETAILED DESCRIPTION:
The protocol was amended in 15 March 2011 to discontinue participants' enrollment and efficacy assessments, and to offer the opportunity for participants already enrolled to continue receiving study treatment for their planned participation in the study. The study had been active in several countries for approximately 1 year, and enrollment had been significantly slower than expected. Thus, the decision was made by the Sponsor to terminate the study since current and projected future enrollment rates would not have provided valuable information in a reasonable timeframe. All clinical efficacy and magnetic resonance imaging (MRI) procedures were removed from the protocol, and safety assessments were to be managed through standard of care activities.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have a diagnosis of relapsing remitting multiple sclerosis (MS) as defined by the revised McDonald Committee criteria (Polman 2005).
2. Must have been treated with a stable regimen of either glatiramer acetate (20 mg per day subcutaneous) or interferon beta-1a (44 mcg 3 times per week subcutaneous) as their principal first therapy for MS for 6 to 18 months prior to randomization. (Note: prior treatment with another MS therapy of ≤ 30 days total duration is not exclusionary [e.g. titration to 44 mcg is allowed]).
3. Have had disease activity within 12 months prior to screening while on therapy; disease activity must be observed after a minimum of 6 months on therapy. Qualifying disease activity is defined as:

   * One or more clinical relapses OR
   * Two or more new MRI lesions (gadolinium [Gd+] and/or T2 hyperintense) For inclusion purposes: (a) a relapse is defined as neurologic signs and/or symptoms documented in the medical record by a neurologist and of sufficient duration to be determined by the Investigator or the Treating Physician as consistent with an MS relapse or (b) MRI activity must be verified by the central reader center.
4. Be naïve to natalizumab.
5. Have a documented Expanded Disability Status Scale (EDSS) score between 0.0 and 5.5, inclusive.

Key Exclusion Criteria:

1. Have a diagnosis of primary progressive, secondary progressive, or progressive relapsing MS (as defined by Lublin and Reingold, 1996). These conditions require the presence of continuous clinical disease worsening over a period of at least 3 months. Patients with these conditions may also have superimposed relapses, but are distinguished from relapsing-remitting patients by the lack of clinically stable periods or clinical improvement.
2. Have known intolerance, contraindication to, or history of non-compliance with, the use of glatiramer acetate or interferon beta-1a.
3. Have had an MS exacerbation (relapse) within 30 days prior to randomization AND/OR the patient has not stabilized from a previous relapse, in the opinion of the Investigator, prior to randomization.
4. The patient is considered by the Investigator to be immunocompromised based on medical history, physical examination, laboratory testing, or due to prior immunosuppressive or immunomodulating treatment.
5. Subjects for whom MRI is contraindicated, i.e., have pacemakers or other contraindicated implanted metal devices, have suffered or are at risk for side effects from gadolinium (Gd), or have claustrophobia that cannot be medically managed.
6. History of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease that would preclude participation in a clinical trial.
7. History of malignant disease, including solid tumors and hematologic malignancies (with the exception of basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
8. Known history of human immunodeficiency virus (HIV).
9. Positive test result for hepatitis C virus (test for hepatitis C virus antibody [HCVAb]) or hepatitis B virus (test for hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb]).
10. History of transplantation or any anti-rejection therapy.
11. History of progressive multifocal leukoencephalopathy (PML).

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (42):
- United States (19):
  - Research Site, Cullman, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Fort Collins, Colorado
  - Research Site, Maitland, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Lexington, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Patchogue, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Round Rock, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Kirkland, Washington
  - Research Site, Morgantown, West Virginia
- Research Site, Fitzroy, Victoria, Australia
- Research Site, Gatineau, Quebec, Canada
- Research Site, Pardubice, Czechia
- Research Site, Tampere, Finland
- Research Site, Strasbourg, Bas-Rhin, France
- Hungary (3):
  - Research Site, Esztergom, Komárom-Esztergom
  - Research Site, Budapest
  - Research Site, Nyíregyháza
- Italy (3):
  - Research Site, Catania, Catania
  - Research Site, Napoli
  - Research Site, Rome
- Research Site, Riga, Latvia
- Poland (3):
  - Research Site, Bialystok, Podlaskie Voivodeship
  - Research Site, Gdansk, Pomeranian Voivodeship
  - Research Site, Lódz, Łódź Voivodeship
- Research Site, Ljubljana, Slovenia
- Spain (6):
  - Research Site, Barcelona, Barcelona
  - Research Site, Alicante
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Seville
- Research Site, Mölndal, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Natalizumab: 300 mg intravenous injection every 4 weeks
Period: Overall Study
Arm/Group | Natalizumab | Interferon Beta-1a | Glatiramer Acetate
Started | 38 | 25 | 21
Dosed With Study Treatment | 36 | 22 | 17
Completed | 0 | 0 | 1
Not Completed | 38 | 25 | 20
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Physician Decision | 2 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 11
Not completed — Withdrawn Due to Study Termination | 27 | 13 | 7
Not completed — Reason Missing | 5 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Natalizumab | Interferon Beta-1a | Glatiramer Acetate | Total
Number analyzed (Participants) | 36 | 22 | 17 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (9.51) | 39.0 (10.0) | 37.6 (13.16) | 37.1 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 16 | 13 | 59
  Male | 6 | 6 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the subject at immediate risk of death (a life-threatening event; however, this does not include an event that, had it occurred in a more severe form, might have caused death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect. An SAE may also have been any other medically important event that, in the opinion of the Investigator, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above. See Adverse Events section below for further details.
Time Frame: up to 108 Weeks
Population: Participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Natalizumab | Interferon Beta-1a | Glatiramer Acetate
Number analyzed (Participants) | 36 | 22 | 17
participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of first dose of study treatment until the final clinic visit (96 weeks); serious adverse events (SAEs) were collected from the time of signed consent to 12 weeks after the last study visit (108 weeks).
Arm/Group | Natalizumab | Interferon Beta-1a | Glatiramer Acetate
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/22 | 0/17
Other Adverse Events (participants affected / at risk) | 19/36 | 12/22 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=36) | Interferon Beta-1a (N=22) | Glatiramer Acetate (N=17)
Meningitis Herpes (Infections and infestations) | 0 | 1 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral Venous Thrombosis (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=36) | Interferon Beta-1a (N=22) | Glatiramer Acetate (N=17)
Urinary Tract Infection (Infections and infestations) | 5 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Gastritis Viral (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 1 | 3 | 5
Headache (Nervous system disorders) | 5 | 2 | 1
Paraesthesia (Nervous system disorders) | 3 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 3 | 0
Migraine (Nervous system disorders) | 2 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0
Loss Of Proprioception (Nervous system disorders) | 0 | 0 | 2
Neuralgia (Nervous system disorders) | 2 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 0 | 1
Orthostatic Tremor (Nervous system disorders) | 0 | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0 | 1
Vitreous Floaters (Eye disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Periodontal Disease (Gastrointestinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 1
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 1
Fatigue (General disorders) | 4 | 2 | 3
Gait Disturbance (General disorders) | 0 | 2 | 1
Pyrexia (General disorders) | 2 | 1 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 2
Influenza Like Illness (General disorders) | 0 | 0 | 1
Injection Site Mass (General disorders) | 0 | 0 | 1
Injection Site Pruritus (General disorders) | 0 | 0 | 1
Injection Site Swelling (General disorders) | 0 | 0 | 1
Heart Rate Increased (Investigations) | 0 | 0 | 1
Vitamin D Decreased (Investigations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Exposure To Toxic Agent (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to early termination of the study and the small size of the study population, there was insufficient power for efficacy and safety analyses. Only serious adverse events were to be captured and reported under the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.